CLINICAL TRIAL: NCT02831387
Title: Randomized, Double-Masked, Parallel Group Study of P-321 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye Disease Assessing Safety and Efficacy Over 28 Days
Brief Title: Evaluation of P-321 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Parion Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-321-202
Record Dates: First submitted 2016-07-01; First posted 2016-07-13 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2017-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.017% P-321 Ophthalmic Solution (Experimental): 0.017% P-321 Ophthalmic Solution TID for 28 days.
  Interventions: Drug: P-321 Ophthalmic Solution
- Placebo (Placebo Comparator): P-321 Ophthalmic Solution Placebo TID for 28 days.
  Interventions: Drug: P-321 Ophthalmic Solution placebo

INTERVENTIONS:
Drug: P-321 Ophthalmic Solution — P-321 Ophthalmic Solution 0.017%
  Other Names: P-321
  Arms: 0.017% P-321 Ophthalmic Solution
Drug: P-321 Ophthalmic Solution placebo — Placebo to match P-321 Ophthalmic Solution
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of treatment with 0.017% P-321 on Dry Eye Symptoms.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-masked, placebo-controlled, parallel group Phase 2b trial designed to evaluate symptoms and signs in subjects with mild to moderate dry eye disease. Eligible patients, will be treated with placebo during 2-week placebo run-in period. Subjects will then be randomly assigned in a double-masked, 1:1 ratio to either 0.017% P-321 Ophthalmic Solution or placebo TID for 28 days. This study is designed to evaluate the changes in symptoms. Safety will be assessed throughout the study by adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Male or female subjects aged 18 to 80 years, inclusive
3. Have a history of dry eye disease (DED) in both eyes
4. Be on stable regimens of other needed medications
5. Have a BCVA of +0.7 or better as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS)
6. Have reported symptoms
7. Have the following signs in at least one eye: Schirmer score without anesthesia of >1 and <10 mm at 5 minutes and staining of conjunctival and corneal areas of the eye.
8. Have normal lid anatomy

Exclusion Criteria:

1. Have undergone refractive eye surgery in the past 12 months
2. Have undergone previous eyelid surgery in either eye (External blepharoplasty not resulting in exposure or abnormal blinking is allowed)
3. Have lid irregularities or deformities
4. Have a history of glaucoma, a history of an elevated lOP within the past year, or an lOP in either eye > 25 mmHg at the Screening Visit (Visit 1)
5. Have any clinically significant, uncontrolled, or unstable medical or surgical conditions that could affect his or her ability to participate
6. Have permanent punctal plugs, punctal occlusion, or history of nasolacrimal duct obstruction. Removable punctal plugs are allowed if they have been used regularly for at least 60 days prior to the screening visit. However, if a plug comes out during the study it must be promptly replaced.
7. Have clinical findings of severe Meibomian Gland Dysfunction (MGD) in the Study Eye
8. Are pregnant or breast feeding
9. Use of any investigational product or device within 28 days prior to the Screening Visit or during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Boyer, Study Director — Parion Sciences
Locations (7):
- United States (7):
  - Sall Research Medical Center, Artesia, California
  - Tauber Eye Center, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Comprehensive Eye Care, Ltd., Washington, Missouri
  - UNC Kittner Eye Center, Chapel Hill, North Carolina
  - Ocular Surface Center, Baylor College of Medicine, Houston, Texas
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Ophthalmic Solution: Subject received Placebo TID administration in both eyes from Visit 2 (Randomization - Treatment Day 1) through the day before Visit 4 (Treatment Day 29)
- 0.017% P-321 Ophthalmic Solution: Subjects received 0.017% P-321 Ophthalmic Solution TID administration in both eyes from Visit 2 (Randomization - Treatment Day 1) through the day before Visit 4 (Treatment Day 29)
Period: Overall Study
Arm/Group | Placebo Ophthalmic Solution | 0.017% P-321 Ophthalmic Solution
Started | 23 | 24
Completed | 22 | 22
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Discontinued due to stock recovery | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Ophthalmic Solution | 0.017% P-321 Ophthalmic Solution | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 17 | 18 | 35
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Visit 2) to Day 29 (Visit 4) in the Subject-reported Dry Eye Symptom Questionnaire.
Description: Dry Eye symptoms were obtained using the Symptom Assessment in Dry Eye (SANDE) questionnaire. The questionnaire utilizes separate Visual Analog Scales (VAS) for the frequency and the Severity of symptoms. The scores range from 0 to 100 where 0 = Rarely or Very Mild, and 100 = All the Time or Very Severe for the Frequency and Severity of the symptoms, respectively. The Global Score as reported in the Primary Outcome is obtained by taking the square root of the product of the frequency score multiplied by the severity score. Negative change from baseline indicates improvement.
Time Frame: Baseline to Day 29
Population: The modified Intent-to-Treat Population (mITT) include all randomized subjects who have at least a baseline and one post-baseline symptom questionnaire part 1 assessment. This is the primary population for efficacy analyses and subjects are analyzed based on their randomized treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Ophthalmic Solution | 0.017% P-321 Ophthalmic Solution
Number analyzed (Participants) | 23 | 24
units on a scale
  Baseline: number analyzed (Participants) | 22 | 23
  Baseline | 58.821 (17.0381) | 59.228 (17.7064)
  Change from Baseline (Visit 2) to Day 29: number analyzed (Participants) | 22 | 22
  Change from Baseline (Visit 2) to Day 29 | -9.197 (24.4776) | -9.989 (12.2523)
Statistical Analysis 1: Comparison: Placebo Ophthalmic Solution vs 0.017% P-321 Ophthalmic Solution; Statistical Analysis 1 for Change From Baseline to Day 29 in the Subject Reported Dry Eye Questionnaire; Test type: Superiority; p = 0.749, Mixed Models Analysis; Mean Difference (Net) = -1.88, 95% CI 2-sided [-13.696 to 9.936]

2. Secondary Outcome: Change From Baseline (Visit 2) to Day 29 in Symptom Frequency Scores
Description: Dry Eye symptom frequency was obtained using the Symptom Assessment in Dry Eye (SANDE) questionnaire. The questionnaire utilizes a 100 mm horizontal Visual Analog Scale (VAS). The scores range from 0 to 100 where 0 = Rarely and 100 = All the Time. A negative change from baseline indicates improvement.
Time Frame: Baseline to Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Ophthalmic Solution | 0.017% P-321 Ophthalmic Solution
Number analyzed (Participants) | 23 | 24
units on a scale
  Baseline: number analyzed (Participants) | 22 | 23
  Baseline | 57.2 (19.58) | 62.3 (17.91)
  Change from Baseline (Visit 2) to Day 29: number analyzed (Participants) | 22 | 22
  Change from Baseline (Visit 2) to Day 29 | -5.3 (25.45) | -12.3 (14.13)
Statistical Analysis 1: Comparison: Placebo Ophthalmic Solution vs 0.017% P-321 Ophthalmic Solution; Statistical Analysis 1 for Change From Baseline (Visit 2) to Day 29 in Frequency Scores; Test type: Superiority; p = 0.267, Mixed Models Analysis; Mean Difference (Net) = -6.6, 95% CI 2-sided [-18.4 to 5.3]

3. Secondary Outcome: Change From Baseline (Visit 2) to Day 29 in Symptom Severity Scores
Description: Dry Eye symptom severity was obtained using the Symptom Assessment in Dry Eye (SANDE) questionnaire. The questionnaire utilizes a 100 mm horizontal Visual Analog Scales (VAS). The scores range from 0 to 100 where 0 = Very Mild and 100 = Very Severe. A negative change from baseline indicates improvement.
Time Frame: Baseline to Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Ophthalmic Solution | 0.017% P-321 Ophthalmic Solution
Number analyzed (Participants) | 23 | 24
units on a scale
  Baseline: number analyzed (Participants) | 22 | 23
  Baseline | 61.1 (15.54) | 56.5 (18.45)
  Change from Baseline (Visit 2) to Day 29: number analyzed (Participants) | 22 | 22
  Change from Baseline (Visit 2) to Day 29 | -13.2 (24.70) | -7.6 (12.88)
Statistical Analysis 1: Comparison: Placebo Ophthalmic Solution vs 0.017% P-321 Ophthalmic Solution; Statistical Analysis 1 for Change From Baseline (Visit 2) to Day 29 in Severity Scores; Test type: Superiority; p = 0.495, Mixed Models Analysis; Mean Difference (Net) = 3.9, 95% CI 2-sided [-7.6 to 15.4]

4. Secondary Outcome: Change From Baseline to Day 29 in Fluorescein Staining of the Cornea.
Description: Corneal staining was performed to grade the corneal epithelial cell injury as measured by fluorescence using slit lamp examination. The staining was graded with the NEI scale. The corneal surface is divided into 5 corneal regions (1, Central; 2, Inferior; 3, Nasal; 4, Temporal; 5, Superior). The scores for each of these 5 regions ranged from 0 to 3 (0=no staining; 1=staining with low density; 2=staining with moderate density; 3=staining with severe density). The total staining score (sum of all regions, maximal score =15) is reported. A negative change from baseline indicates improvement.
Time Frame: Baseline to Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Ophthalmic Solution | 0.017% P-321 Ophthalmic Solution
Number analyzed (Participants) | 23 | 24
units on a scale
  Baseline: number analyzed (Participants) | 22 | 23
  Baseline | 5.8 (1.31) | 6.3 (1.58)
  Change from Baseline (Visit 2) to Day 29: number analyzed (Participants) | 22 | 22
  Change from Baseline (Visit 2) to Day 29 | -1.2 (2.4) | -0.7 (2.68)
Statistical Analysis 1: Comparison: Placebo Ophthalmic Solution vs 0.017% P-321 Ophthalmic Solution; Statistical Analysis 1 for Change From Baseline to Day 29 in Fluorescein Staining of the Cornea; Test type: Superiority; p = 0.316, Mixed Models Analysis; Mean Difference (Net) = 0.6, 95% CI 2-sided [-0.6 to 1.9]

5. Secondary Outcome: Change From Baseline to Day 29 in Lissamine Green Staining of the Conjunctiva.
Description: Conjunctival staining was performed to grade the conjunctival epithelial cell injury as measured by Lissamine Green using slit-lamp examination. The staining was graded with the NEI scale. The bulbar conjunctival surface is divided into 6 regions (1, Temporal; 2 Temporal Superior; 3, Temporal Inferior; 4, Nasal Superior; 5, Nasal Inferior; 6, Nasal). The scores for each of these 6 regions ranged from 0 to 3 (0=no staining; 1=staining with low density; 2=staining with moderate density; 3=staining with severe density). The total staining score (sum of all regions, maximal score =18) is reported. A negative change from baseline indicates improvement.
Time Frame: Baseline to Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Ophthalmic Solution | 0.017% P-321 Ophthalmic Solution
Number analyzed (Participants) | 23 | 24
units on a scale
  Baseline: number analyzed (Participants) | 22 | 23
  Baseline | 7.6 (1.73) | 7.1 (1.79)
  Change from Baseline (Visit 2) to Day 29: number analyzed (Participants) | 22 | 22
  Change from Baseline (Visit 2) to Day 29 | -0.3 (3.41) | -0.2 (3.78)
Statistical Analysis 1: Comparison: Placebo Ophthalmic Solution vs 0.017% P-321 Ophthalmic Solution; Statistical Analysis 1 for Change From Baseline to Day 29 in Lissamine Green Staining of the Conjunctiva; Test type: Superiority; p = 0.823, Mixed Models Analysis; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.9 to 1.5]

6. Secondary Outcome: Number of Participants With at Least 20% Improvement in Symptoms From Baseline to Day 29
Description: Improvement in symptoms was evaluated using the Symptom Assessment in Dry Eye (SANDE) questionnaire. The questionnaire utilizes separate Visual Analog Scales (VAS) for the frequency and the Severity of symptoms. The scores range from 0 to 100 where 0 = Rarely or Very Mild, and 100 = All the Time or Very Severe for the Frequency and Severity of the symptoms, respectively. The Global Score is obtained by taking the square root of the product of the frequency score multiplied by the severity score. Lower scores indicate improvement in symptoms.
Time Frame: Baseline to Day 29
Population: The modified Intent-to-Treat Population (mITT) include all randomized subjects who have at least a baseline and one post-baseline symptom questionnaire part 1 assessment. For this outcome, only participants that completed the treatment were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Ophthalmic Solution | 0.017% P-321 Ophthalmic Solution
Number analyzed (Participants) | 22 | 22
Participants | 8 | 11
Statistical Analysis 1: Comparison: Placebo Ophthalmic Solution vs 0.017% P-321 Ophthalmic Solution; Statistical Analysis 1 for the Number of participants with at least 20% improvement in symptoms from baseline to Day 29; Test type: Superiority; Odds Ratio (OR) = 1.923, 95% CI 2-sided [0.515 to 7.184]

7. Secondary Outcome: Change From Baseline (Visit 2) to Day 15 (Visit 3) in the Subject-reported Dry Eye Symptom Score.
Description: Dry Eye symptoms were obtained using the Symptom Assessment in Dry Eye (SANDE) questionnaire. The questionnaire utilizes separate Visual Analog Scales (VAS) for the frequency and the Severity of symptoms. The scores range from 0 to 100 where 0 = Rarely or Very Mild, and 100 = All the Time or Very Severe for the Frequency and Severity of the symptoms, respectively. The Global Score as reported in the Primary Outcome is obtained by taking the square root of the product of the frequency score multiplied by the severity score. A negative change from baseline indicates improvement.
Time Frame: Baseline to Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Ophthalmic Solution | 0.017% P-321 Ophthalmic Solution
Number analyzed (Participants) | 23 | 24
units on a scale
  Baseline: number analyzed (Participants) | 22 | 23
  Baseline | 58.821 (17.0381) | 59.228 (17.7064)
  Change from Baseline (V2) to Day 15 (V3): number analyzed (Participants) | 22 | 23
  Change from Baseline (V2) to Day 15 (V3) | -4.759 (16.0865) | -2.985 (16.2819)
Statistical Analysis 1: Comparison: Placebo Ophthalmic Solution vs 0.017% P-321 Ophthalmic Solution; Statistical Analysis 1 for Change From Baseline (Visit 2) to Day 15 (Visit 3) in the Subject-reported Dry Eye Symptom Score; Test type: Superiority; p = 0.723, Mixed Models Analysis; Mean Difference (Net) = 1.666, 95% CI 2-sided [-7.759 to 11.092]

ADVERSE EVENTS:
Time Frame: 29 days
Description: An AE was defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product, which did not necessarily have to have a causal relationship with this treatment. A treatment-emergent AE (TEAE) was an AE that either commenced following initiation of study treatment or was present prior to study treatment but increased in frequency or severity following initiation of study treatment.
Arm/Group | 0.017% P-321 Ophthalmic Solution | Placebo Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 4/24 | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.017% P-321 Ophthalmic Solution (N=24) | Placebo Ophthalmic Solution (N=23)
Conjunctival disorders (Eye disorders) | 1 (1) | 0 (0)
Eyelid Oedema (Eye disorders) | 1 (2) | 0 (0)
Instillation Site Pain (Eye disorders) | 0 (0) | 1 (1)
Fatigue (Eye disorders) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Eye disorders) | 1 (1) | 0 (0)
Muscle Strain (Eye disorders) | 0 (0) | 1 (1)
Dysgeusia (Eye disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator may publish or present the results based on data generated at their Institution, provided that: (a) Sponsor publishes the results from all sites participating in the Study; (b) Institution receives notification from Sponsor that publication of the multi-site results is no longer planned; or (c) eighteen (18) months following the close of study, whichever occurs first.

DOCUMENTS (2):
  • Study Protocol (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT02831387/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT02831387/SAP_001.pdf